CLINICAL TRIAL: NCT06920043
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled Study of Efimosfermin Alfa in Participants With Biopsy-confirmed Cirrhosis (Compensated) Due to Metabolic Dysfunction-associated Steatohepatitis (MASH)
Brief Title: A Study of Efimosfermin Alfa in Participants With Biopsy-confirmed Cirrhosis (Compensated) Due to MASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 306301 (BOS-580-202)
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis
Keywords: Fibroblast growth factor; Stage 4 fibrosis; Compensated Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efimosfermin (Dose 1) (Experimental): Participants will receive efimosfermin (Dose 1) once every 4 weeks (Q4W).
  Interventions: Drug: Efimosfermin
- Efimosfermin (Dose 2) (Experimental): Participants will receive efimosfermin (Dose 2) Q4W.
  Interventions: Drug: Efimosfermin
- Placebo (Placebo Comparator): Participants will receive placebo Q4W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efimosfermin — Efimosfermin will be administered as a subcutaneous injection.
  Other Names: BOS-580
  Arms: Efimosfermin (Dose 1); Efimosfermin (Dose 2)
Drug: Placebo — Placebo will be administered as a subcutaneous injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, preliminary efficacy, and pharmacokinetics (PK) of efimosfermin in participants with metabolic dysfunction associated steatohepatitis (MASH) and compensated cirrhosis consistent with stage F4 fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form (ICF)
* Age 18 through 75 years at enrollment
* History or presence of 2 or more of the 5 components of metabolic syndrome
* Liver biopsy confirmation of MASH consistent with stage F4 fibrosis
* Other inclusion criteria may apply.

Exclusion Criteria:

* Individuals with chronic liver disease from other causes, or any history or evidence of decompensated liver disease
* History of type 1 diabetes
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥5 × the upper limit of normal (ULN)
* Other exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | From Day 1 to 100 weeks
  To assess the effects of efimosfermin on safety and tolerability.

SECONDARY OUTCOMES:
Serum concentrations of efimosfermin | Up to Week 21
  To assess the steady-state PK of efimosfermin.
Maximum serum drug concentration (Cmax) of efimosfermin | Up to Week 21
  To assess the steady-state PK of efimosfermin.
Area under the serum concentration-time curve (AUC) of efimosfermin | Up to Week 21
  To assess the steady-state PK of efimosfermin.
Average serum drug concentration (Cavg) of efimosfermin | Up to Week 21
  To assess the steady-state PK of efimosfermin.
Concentration of study drug at the end of the dosing interval (Ctrough) of efimosfermin | Up to Week 21
  To assess the steady-state PK of efimosfermin.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - Arizona Liver Health - Peoria, Peoria, Arizona
  - The Institute for Liver Health II LLC dba Arizona Liver Health - Tucson, Tucson, Arizona
  - Fresno Clinical Research Center, Fresno, California
  - OM Research LLC, Lancaster, California
  - Knowledge Research Center, Orange, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - Santa Maria Gastroenterology Center, Santa Maria, California
  - ClinCloud Research - Maitland, Maitland, Florida
  - ClinCloud Research - Viera, Melbourne, Florida
  - Advanced Clinical Research of Miami, Miami, Florida
  - Centricity Research - Columbus, Columbus, Georgia
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - Mercy Medical Center - Baltimore, Maryland, Baltimore, Maryland
  - Gastrointestinal Associates and Endoscopy Center, PA - Flowood, Flowood, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - IMA Clinical Research - Austin, TX, Austin, Texas
  - American Research Corporation - Austin, TX, Austin, Texas
  - Pinnacle Clinical Research - Austin, TX, Austin, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Pinnacle Clinical Research - Georgetown, Georgetown, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Research Institute - Texas Medical Center, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - LinQ Research, LLC, Katy, Texas
  - Houston Research Institute - Pasadena, Pasadena, Texas
  - American Research Corporation - San Antonio, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Velocity Clinical Research - Waco, Waco, Texas
  - Richmond Institute for Veterans Research, Richmond, Virginia
  - GI Alliance - Washington Gastroenterology, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No